CLINICAL TRIAL: NCT01998503
Title: Induction Therapy With Bortezomib and Dexamethasone Followed by Autologous Stem Cell Transplantation Versus Autologous Stem Cell Transplantation Alone in the Treatment of AL Amyloidosis
Brief Title: Bortezomib and Dexamethasone Followed by ASCT Compared With ASCT Alone in Treating Patients With AL Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0703
Record Dates: First submitted 2013-11-15; First posted 2013-11-29 (Estimated); Last update posted 2013-11-29 (Estimated); Status verified 2013-11

CONDITIONS: Amyloidosis
Keywords: AL amyloidosis; bortezomib; autologous stem cell transplantation
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Dexamethasone; Filgrastim; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BD induction followed by ASCT (Active Comparator): The BD regimen included bortezomib 1.3 mg/m2 i.v. and dexamethasone 40 mg p.o. on days 1, 4, 8 and 11 of the 21 day cycle. This process was repeated for 2 cycles. After two cycles of BD therapy, the collection of peripheral blood stem cells (PBSC) should be completed within 4 weeks. Patients receive filgrastim (G-CSF) on days 1 to 5 and undergo autologous hematopoietic stem cell (HSC) collection. Patients will receive ASCT therapy in 8 weeks after collection of PBSC (Recorded as day 0), while melphalan (day -2) with a dose of 140 or 200 mg/m2 (choosing a dose according to the degree of risk for patients). Melphalan will be administered by central venous catheter.
  Interventions: Drug: Bortezomib; Drug: dexamethasone; Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation (ASCT); Drug: Melphalan
- ASCT alone (Experimental): the patients who assigned to this arm will receive ASCT alone as an initial treatment. At first, patients receive the collection of peripheral blood stem cells (PBSC), Patients receive filgrastim (G-CSF) on days 1 to 5 and undergo autologous hematopoietic stem cell (HSC) collection. After then patients will receive ASCT therapy in 8 weeks after collection of PBSC (Recorded as day 0), while melphalan (day -2) with a dose of 140 or 200 mg/m2 (choosing a dose according to the degree of risk for patients). Melphalan will be administered by central venous catheter.
  Interventions: Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation (ASCT); Drug: Melphalan

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade
  Arms: BD induction followed by ASCT
Drug: dexamethasone — Given orally
  Arms: BD induction followed by ASCT
Biological: filgrastim — Given subcutaneous
Procedure: autologous hematopoietic stem cell transplantation (ASCT) — Given on day 0
Drug: Melphalan

SUMMARY:
This randomized phase III trial is studying the side effects and how well giving induction therapy with bortezomib and dexamethasone followed by autologous stem cell transplantation (ASCT) compared with ASCT alone in treating patients with newly diagnosed renal AL amyloidosis. In this prospective, randomized control study, patients with newly diagnosed AL amyloidosis who met the criteria for ASCT were randomized to receive 2 cycles of BD as induction therapy followed by ASCT (BD+ASCT) (arm 1) or to receive ASCT alone as an initial treatment (arm 2). Hematologic and organ responses were evaluated every 3 months after ASCT. All the patients should be followed up for 12 months.

DETAILED DESCRIPTION:
Arm 1: The BD regimen included bortezomib 1.3 mg/m2 i.v. and dexamethasone 40 mg p.o. on days 1, 4, 8 and 11 of the 21 day cycle. This process was repeated for 2 cycles. After two cycles of BD therapy, the collection of peripheral blood stem cells (PBSC) should be completed within 4 weeks. Recommended dose of drug is as follows: granulocyte colony-stimulating factor (G-CSF) 5-10ug/kg on days 1-5 will be given, then peripheral blood stem cells will be collected on days 5-6 for 2×10^6 CD34+ cells /kg. Patients will receive ASCT therapy in 8 weeks after collection of PBSC (Recorded as day 0), while melphalan (day -2) with a dose of 140 or 200 mg/m2 (choosing a dose according to the degree of risk for patients). Melphalan will be administered by central venous catheter.

Arm 2: the patients who assigned to arm 2 will receive ASCT alone as an initial treatment. The process of ASCT is as same as arm 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AL amyloidosis
* Abnormal M protein or free light chain detected in serum and/or urine
* ECOG score 0-2 points
* No absolute neutrophil count of ANC less than or equal to 1000 within 14 days before enrollment
* No platelet count of less than or equal to 50K within 14 days before enrollment
* Serum bilirubin must lower than 2.0 mg/dl within 14 days before enrollment
* Serum creatinine must lower than 2.0 mg/dl within 14 days before enrollment
* Must have LVEF at least 45% by ECHO within 14 days of enrollment
* Pulmonary Function Tests must show DLCO at least 50%

Exclusion Criteria:

* Subjects have received or are currently receiving systematic treatment with steroids (not including an emergent short-term use of steroids before randomization up to 4 days, maximum dose of 40mg/d)
* Pregnant and breastfeeding women, delivery term women or unwilling to take birth control measures during the study
* Subjects suffering from multiple myeloma
* Grade 2 or more than grade 2 peripheral neuropathy or neuropathic pain according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3
* Known or suspected hypersensitivity to dexamethasone, bortezomib, mannitol, boron, or heparin (if use catheters)
* Subjects suffering from uncontrolled or severe cardiovascular disease, including myocardial infarction, class III-IV heart failure defined by New York Heart Association (NYHA), uncontrolled angina, clinical significant pericardial disease or cardiac amyloidosis (Other contraindications are not suitable for transplant patients) within 6 months before enrollment
* Subjects suffering from serious physical disease and mental illnesses which may interfere the study
* Subjects receiving other pilot study or treatment within 4 weeks before enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with hematologic complete response between BD+ASCT arm and ASCT alone arm in the treatment of AL amyloidosis | 12 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 12 months
Number of participants with organ responses between BD+ASCT arm and ASCT alone arm in the treatment of AL amyloidosis | 12 months
Overall survival | 24 months
Progression free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Huang X, Wang Q, Chen W, Zeng C, Chen Z, Gong D, Zhang H, Liu Z. Induction therapy with bortezomib and dexamethasone followed by autologous stem cell transplantation versus autologous stem cell transplantation alone in the treatment of renal AL amyloidosis: a randomized controlled trial. BMC Med. 2014 Jan 6;12:2. doi: 10.1186/1741-7015-12-2. PMID 24386911